CLINICAL TRIAL: NCT03066167
Title: Validation of Instruments Used for Assessment of Dysphagia in Patients With Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other); The Göteborg Medical Society, Sweden (Unknown)
Responsible Party: Sponsor
Other Study IDs: janpe4(2)
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Dysphagia, Esophageal; Esophageal Cancer
Keywords: Cancer of the gastro-esophageal junction; Watson score; Ogilvie score; Goldschmid score; Validation; Quality of Life
MeSH Terms: conditions — Deglutition Disorders; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients: Patients with oesophageal cancer and dysphagia
  Interventions: Other: Validation of different dysphagia scores
- Controls: Healthy Controls with no known dysphagia
  Interventions: Other: Validation of different dysphagia scores

INTERVENTIONS:
Other: Validation of different dysphagia scores
  Other Names: Validation to the Swedish language

SUMMARY:
This study validates 3 well known dysphagia scores for dysphagia due to malignancies of the oesophagus and gastro-oesophageal junction and to the Swedish language.

DETAILED DESCRIPTION:
In the present study, our aim was to firstly, validate 3 commonly used scales for use in patients with dysphagia due to malignancy, and secondly, to validate them in the Swedish language. The 3 scales were: The Watson dysphagia scale, which was developed in studies on surgical treatment of reflux disease. It consists of questions about food with 9 different viscosity and solidity and the patient answer if they have problems with a specific food: never, sometimes or always when ingesting this. The scores are added and provides a range of 0-45 where 45 is the worst possible dysphagia. The Ogilvie score is a 5-graded scale 0-4 where 4 is total inability to swallow. The Goldschmid score is graded from 0-5 where 0 is inability to swallow and 5 is normal function. QoL was measured with validated instruments originating from the European Organization for Research and Treatment of Cancer (EORTC), which has a generic instrument that measures global QoL in patients with cancer (QLQ-C30) and a more symptom-specific instrument that is developed for cancer in the oesophagus and stomach (QLQ-OG25). These are well known, validated instruments that also have normal reference values for the healthy population. The symptom specific instrument QLQ-OG25 includes a dysphagia module consisting of 3 questions which is validated to malignant disease and food intake with the help of expert groups and deep interviews with patients.

ELIGIBILITY:
Inclusion Criteria:

* Cancer in the gastro-esophageal junction or in the esophagus
* Dysphagia
* Ability to fill in the questionnaires
* Written acceptance of the informed consent

Exclusion Criteria:

* Not for-filling inclusion criteria
* No consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cancer in the oesophagus and as Controls, healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Validation of dysphagia scores | 10-14 days
Translation of scores to the Swedish language | 10-14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Department, Sahlgrenska University Hospital, Gothenburg, Västra Götalandsregionen, Sweden

IPD SHARING:
Plan to Share IPD: No